CLINICAL TRIAL: NCT02747784
Title: Randomized Evaluation to Assess Cognitive Training for the Prevention of Post-operative Cognitive Decline (REACT) - a Pilot Study
Brief Title: Evaluation to Assess Cognitive Training for the Prevention of Post-operative Cognitive Decline
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine, Campus Virchow - Klinikum (CVK)/Campus Charité Mitte (CCM), Charité - University Medicine Berlin, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REACT
Record Dates: First submitted 2016-03-30; First posted 2016-04-22 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Dysfunction
Keywords: cognitive dysfunction; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group experimental (Experimental): 24 female patients aged 18 years or older undergoing urogynecological or breast cancer surgery; the patients are recommended to perform the RehaCom® training modules 'Topological Memory (MEMO)' and 'Divided Attention 2 (GEA2)' daily during inpatient hospital stay, and at least three times a week for 30 to 60 minutes until month 3.
  Interventions: Behavioral: Cognitive training program RehaCom®
- Study group active comparator (Active Comparator): 24 female patients aged 18 years or older undergoing urogynecological or breast cancer surgery; the patients are recommended to perform the RehaCom® training modules 'Topological Memory (MEMO)' and 'Working memory (WOME)' daily during inpatient hospital stay, and at least three times a week for 30 to 60 minutes until month 3.
  Interventions: Behavioral: Cognitive training program RehaCom®
- Control group (No Intervention): 48 female control subjects aged 18 years or older (24 without surgery, 24 with urogynecological or breast cancer surgery) with a similar health status and age as the study group patients (similar distribution in the American Society of Anaesthesiologists physical status classification and relevant co-morbidities, e.g. diabetes, coronary artery disease, hypertension and hyperlipidemia). The patients are analyzed to correct for learning effects of the cognitive assessment testings in the study groups.

INTERVENTIONS:
Behavioral: Cognitive training program RehaCom® — Cognitive training program RehaCom®
  Arms: Study group active comparator; Study group experimental

SUMMARY:
The purpose of this open, monocentric randomized, parallel-group, controlled trial is to compare two different computer-based cognitive training programs regarding the efficacy to prevent the 3-months incidence of postoperative cognitive dysfunction in female patients after elective urogynecological or breast cancer surgery.

DETAILED DESCRIPTION:
The REACT trial has been designed as a feasibility study to investigate the impact of pre-, peri-, and postoperative computerized cognitive trainings on the incidence of postoperative cognitive dysfunction. Two different study groups (training programs) will be compared. Each group consists of two training modules of the validated computer based training program of cognitive functioning called RehaCom®. The experimental group consists of the modules 'Topological Memory (MEMO)' and 'Divided Attention 2 (GEA2)'. The active comparator group consists of the modules 'Topological Memory (MEMO)' and 'Working memory (WOME)'. 48 surgical patients undergoing elective urogynecological or breast cancer surgery will preoperatively be randomly assigned to one of two study groups. Before starting the training, patients will complete a neuropsychological test battery comprising the cognitive tests to measure POCD. The tests will be assessed at preoperative baseline visit and at 3-months follow-up. In order to correct change in cognitive performance for practice effects, a group of 24 female surgical control subjects will also prospectively be tested with the cognitive test battery at baseline and 3-months follow-up. The control subjects will be matched to the 2 study groups regarding health status, surgery and age, but will neither undergo the computerized cognitive training program RehaCom®. Further, 24 female control subjects are included from the POCD-Register (EA1/104/16) and will be matched to the 2 study groups as well.

After baseline assessment, the study group patients will be taught to use the training program RehaCom®, and training should start preoperatively as early as possible. The patients are recommended to perform the training daily during inpatient hospital stay, and at least three times a week for 30 to 60 minutes until month 3.

The neuropsychological assessment will be performed at preoperative baseline and at three-months follow-up. Postoperative cognitive dysfunction (POCD) will be classified using the dichotomous approach established by Rasmussen et al in the International Study on postoperative cognitive deficits (ISPOCD) (Rasmussen et al. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89.) This calculation method defines POCD as a reliable change in pre- and postoperative cognitive performance (difference scores) of each individual in the surgical patients cohort as compared to the changes in a non-surgical control group (reliable change index in either a composite score including cognitive test parameters from all tests in the cognitive test battery or in at least two of the chosen cognitive test parameters).

Secondary outcome measures of this trial comprise structural and functional MRI measures, Electroencephalogram simultaneous with fMRI, intraoperative cerebral oximetry and neuromonitoring, delirium, pain, sleep quality, postoperative complications, frailty, psychological distress, quality of life, training performance and evaluation of the training.

ELIGIBILITY:
Study groups

Inclusion Criteria:

* Pilot study: Female patients undergoing urogynecological or breast cancer surgery, screened at the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany
* Age 18 years or older
* Montreal Cognitive Assessment Score (MOCA) > 25
* Patient has access to Personal computer or Laptop with system software Windows XP Service Pack 3 (or newer); tablets or smart phones cannot by used.
* Written informed consent to participate after having been properly instructed
* Written informed consent that accidental clinically relevant diagnostic findings of MRI assessment are reported to the general practitioner of the patient
* Sufficient health insurance to cover additional diagnostic assessments in case of an accidental clinically relevant diagnostic finding of MRI assessment

Exclusion Criteria:

* Apparent dementia
* Lacking willingness to take part in the study, or to have relevant study data collected, saved and analyzed for the purpose of the study
* Lacking willingness to be contacted by telephone or mail.
* Accommodation in an institution due to an official or judicial order
* Insufficient knowledge of German language
* Members of the hospital staff
* Admitted in police custody
* Homelessness or other conditions that disable reachability for postoperative assessment by post or telephone
* Illiteracy
* Severe hearing impairment that affects the neuropsychological testing.
* Severe visual impairment that affects the neuropsychological testing.
* Participation in other prospective clinical interventional trials
* Daltonism
* Contra-indications against MRI assessment (claustrophobia, metallic implants, cardiac pacemaker, tatoos)
* Motor impairment that affects the use of a computer
* Regular use of psychotropic drugs (including sleep-inducing drugs and benzodiazepines) and substances which affect cognitive performance Control group

Inclusion Criteria:

24 female surgical control subjects from the POCD Register (EA1/104/169) and 24 female non-surgical control subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients undergoing urogynecological or breast cancer surgery, screened at the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany
Enrollment: 19 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (POCD) | Up to 3 months
  Cognitive functioning will be measured with a battery of computerized neuropsychological tests, non-computerized and computer-based tests from the Cambridge Neuropsychological Test Automated Battery [CANTAB®]

SECONDARY OUTCOMES:
Divided attention | Up to 3 months
  Divided attention will be measured in the pilot study with the Test of Attentional Performance - Mobility version (TAP-M), subtests divided attention and distractibility.
Incidence of postoperative delirium | Up to 7 days
  Postoperative delirium rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and Chart Review
Intraoperative depth of sedation | At time of surgery
  Intraoperative depth of sedation will be monitored in the pilot study with changes in the pattern off EEG-raw data measured with the Masimo SedLine® brain function monitoring for Root®.
Depth of sedation on the Intensive Care Unit | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Depth of sedation will be measured in the pilot study with the Richmond Agitation Sedation Scale (RASS)
Intraoperative cerebral oximetry | At time of surgery
  Intraoperative cerebral oximetry will be measured in the pilot study by near-infrared spectroscopy (NIRS) developed for the Masimo Root® monitor.
Quality of sleep | Up to 3 months
  Quality of sleep will be measured with the Insomnia Severity Index (ISI)
Anxiety | Up to hospital discharge, an expected average of 7 days
  Perioperative anxiety will be measured with the Faces Anxiety Scale (FAS) during hospital stay.
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Evaluation of the cognitive training program RehaCom® by patient | Up to 3 months
  The evaluation will be measured with single items concerning patients' subjective rating of the quality of the training program, at least once during the week
Performance of cognitive training units of the program RehaCom® | Up to 3 months
  Data will be saved automatically by the computerized training program. The training performance will be measured as the highest level a patient has reached per training module, as well as number of mistakes within each level.
Duration of the cognitive training of the program RehaCom® | Up to 3 months
  Data will be saved automatically by the computerized training program. Duration will be measured as minutes per session and total sum of minutes of all sessions.
Frequency of the cognitive training of the program RehaCom® | Up to 3 months
  Data will be saved automatically by the computerized training program. Frequency will be measured as number of sessions and number of weeks with at least 1 session per week.
MRI assessment | Up to 3 months
  Functional MRI: Changes in neural activations in temporal and fronto-parietal brain regions during recognition in a face-name association task at baseline and three months after baseline assessment
MRI assessment | Up to 3 months
  Structural MRI: Changes in gray and white matter.
MRI assessment | Up to 3 months
  Functional MRI: Changes in neural activations in temporal and fronto-parietal brain regions during memory encoding at baseline and three months after baseline assessment
Barthel Activities of Daily Living (ADL) Index | Up to 3 months
  Functional Status will be assessed with the Barthel Activities of Daily Living (ADL) Index
Instrumented Activities of Daily Living (IADL) | Up to 3 months
  Functional Status will be assessed with the Instrumented Activities of Daily Living (IADL) scores
Frailty | Up to 3 months
  Frailty will be measured by modified Fried's criteria (Physical Frailty Phenotype)
Generalized anxiety | Up to 3 months
Depression | Up to 3 months
  Depression will be measured with the Patient Health Questionnaire 9-Item Scale (PHQ-9).
Quality of life | Up to 3 months
  Quality of life will be measured with a standardized instrument for use as a measure of health outcome EQ-5D
Routine laboratory | Up to hospital discharge, an expected average of 7 days
  No additional blood samples will be taken in the pilot study
Organ dysfunctions | Up to hospital discharge, an expected average of 7 days
  Organ dysfunctions are evaluated according to the Clavien-Dindo classification of surgical complications
Mortality | Up to three months
  Mortality is evaluated in the pilot study
Postoperative pain | Up to 3 months
  Postoperative pain will be measured with the Numeric Rating Scale (NRS-V) and validated scores
Mild cognitive impairment | Up to 3 months
  Mild cognitive impairment will be measured by impaired performance in neuropsychological testing (neurocognitive test battery), level of functionality (ADL, IADL) and self report on cognitive impairment (Metamemory and FEDA questionnaire) and related to performance in the MOCA cognitive screening tool.
Timed up and go test | Up to 3 months
Continence | Up to 3 months
  Measured by Deutscher Beckenboden-Fragebogen
Self report on cognitive deficits | Up to 3 months
  Fragebogen erlebter Defizite der Aufmerksamkeit (FEDA)
Metamemory | Up to 3 months
  Multifactorial Memory Questionnaire
Fatigue | Up to 3 months
  2 questions
Assessment on cognitive deficits by Proxy (IQCODE) | Up to 3 months
  Informant Questionnaire on Cognitive Decline in the Elderly
BIA (Bio-Impedanz-Analysis) | Up to 3 months
MNA Mini nutritional assessment-MNA short form) | Up to 3 months
Risk factors of dementia | Up to 3 months
  Risk factors of dementia are analysed by blood levels of APOE-4, BDNF, Kynurenine, Zonulin, Endocan and Tryptophan
Pro- und anti-inflammatory cytokines | Up to 3 months
micro-RNA | Up to 3 months

OTHER OUTCOMES:
Medication history | From date of inclusion until the date of the beginning of surgery, assessed up to 1 week
Diabetic "yes"/"no" | From date of inclusion until the date of the beginning of surgery, assessed up to 1 week day
Mehrfachwahl-Wortschatztest Form A | From date of inclusion until the date of the beginning of surgery, assessed up to 1 week
  Intelligence is assessed using a multiple-choice vocabulary test (MWTA; Mehrfachwahl-Wortschatztest Form A). This test measures crystallized intelligence, which is the ability to use skill, knowledge, and experience and which relies on information from long-term memory.
Falls within last year | From date of inclusion until the date of the beginning of surgery, assessed up to 1 week day
Charlson Comorbidity index | From date of inclusion until the date of the beginning of surgery, assessed up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462